CLINICAL TRIAL: NCT07305675
Title: Effectiveness of a rhGM-CSF-containing Gel on Promoting Recovery After 1927-nm Fractional Thulium Fiber Laser Treatment of Atrophic Acne Scars: a Prospective, Randomized, Split-face, and Evaluator-blinded Clinical Trial
Brief Title: Effectiveness of a rhGM-CSF-containing Gel on Promoting Recovery After 1927-nm Fractional Thulium Fiber Laser Treatment of Atrophic Acne Scars.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Weihui Zeng, Professor, Second Affiliated Hospital of Xi'an Jiaotong University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024220
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Acne Scars - Atrophic; Wound Healing
Keywords: Acne Scars; fractional thulium fiber laser; Granulocyte-macrophage colony-stimulating factor; Acute wound healing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rhGM-CSF side (Experimental): We applied rhGM-CSF-containing gel (Changchun GeneScience Pharmaceutical Corporation Ltd, China) twice daily (100mg/(cm2*d)) for 7 days after 1927-nm TFL therapy.
  Interventions: Drug: rhGM-CSF-containing gel; Device: 1927-nm TFL
- Control Side (Other): No intervention after 1927-nm TFL therapy
  Interventions: Device: 1927-nm TFL

INTERVENTIONS:
Drug: rhGM-CSF-containing gel — rhGM-CSF side was applied recombinant human granulocyte-macrophage colony-stimulating factor-containing gel twice daily (100mg/(cm2*d)) for 7 days from baseline.
  Arms: rhGM-CSF side
Device: 1927-nm TFL — All enrolled patients received once 1927-nm fractional thulium fiber laser (WONTECH, Lavieen, South Korea) treatment on both sides of the face at baseline.

SUMMARY:
Atrophic acne scars (AAS) is one of the most common skin sequelae following acne vulgaris. Fractional laser has shown great therapeutic potential in recent years, while there is no standard of wound care after laser resurfacing. Granulocyte-macrophage colony-stimulating factor (GM-CSF) is a multifunctional cytokine, and has shown its value in many other acute wounds healing. In the present study, we investigated the efficacy and safety of topical recombinant human GM-CSF combined with 1927-nm fractional thulium fiber laser (TFL) in AAS treatment.

DETAILED DESCRIPTION:
Acne vulgaris is a prevalent chronic inflammatory skin disorder affecting approximately 9% of the global population, with 3-7% of patients developing scarring. Among these, atrophic acne scars (AAS) are the most common subtype, exerting profound aesthetic and psychological burdens that substantially impair patients' quality of life.

The 1927-nm fractional thulium fiber laser (TFL) has emerged as a leading treatment for AAS due to its ability to induce controlled microthermal injury in the superficial dermis, stimulating collagen remodeling and dermal regeneration. Its favorable safety profile-characterized by minimal tissue trauma, rapid recovery, and a low risk of post-inflammatory hyperpigmentation (PIH)-supports its clinical utility. Nonetheless, during the treatment of AAS, the ablative energy generated by the laser inevitably leads to disruption of the epidermal barrier and thermal injury, often resulting in erythema, exudation, crusting, or pigmentation changes during recovery.

Cutaneous wound healing is a multifactorial biological process involving coordinated inflammation, proliferation, and tissue remodeling. Cytokines are essential mediators in this cascade, orchestrating angiogenesis, fibroblast activation, and epithelial regeneration to restore barrier integrity. In the context of post-laser skin wound healing, cytokine-based interventions such as epidermal growth factor (EGF) and fibroblast growth factor (FGF) have demonstrated efficacy in enhancing re-epithelialization and reducing adverse sequelae.

Granulocyte-macrophage colony-stimulating factor (GM-CSF) is a multifunctional cytokine secreted by keratinocytes, macrophages, and T lymphocytes that promotes fibroblast proliferation, keratinocyte migration, angiogenesis, and granulation tissue formation. Emerging research suggests its efficacy in wound healing. Distinct from EGF and FGF, GM-CSF also modulates local inflammation, improves microcirculation, and reduces infection risk, thereby optimizing the immune and metabolic milieu for cutaneous repair. Topical GM-CSF formulations have shown promising outcomes in chronic ulcers, radiation dermatitis and burns, accelerating wound closure and minimizing scar formation. However, evidence regarding its efficacy in laser-induced skin injury remains scarce.

This study represents the first investigation of recombinant human GM-CSF (rhGM-CSF) gel as an adjunctive therapy following 1927-nm TFL treatment for atrophic acne scars. We aimed to evaluate its efficacy in promoting postoperative wound healing and restoring skin barrier function, as well as its clinical value in reducing inflammation, enhancing patient comfort, shortening recovery time, and preventing hyperpigmentation. These findings may provide a theoretical basis for developing optimized, cytokine-assisted post-laser repair strategies in aesthetic dermatology.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with atrophic acne scars with essentially symmetric bilateral facial lesion areas, and a Global Scarring Severity (GSS) scale score of Grade 2 or 3 (qualitative assessment);
* Patients with normal cognitive function and mental status;
* Patients with adequate communication ability;
* Patients who voluntarily participate in the split-face controlled study and provide written informed consent.

Exclusion Criteria:

* Having received systemic medications, dermabrasion, or laser therapy within the past 3 months;
* Females who are pregnant, lactating, or planning to become pregnant;
* Presence of severe systemic diseases;
* Psychiatric disorders or impaired capacity for self-care;
* Photosensitivity or having taken photosensitizing medications within the past month;
* Atopic diathesis or history of severe allergic reactions;
* History of skin exposure to intense sunlight within the past month;
* History of keloid formation;
* Presence of active skin tumors or infections;
* Subjects allergic to rhGM-CSF gel or similar products;
* Other subjects deemed ineligible for the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
IGA score | 0,1,2,3,4,5,6,7 days
  The IGA score can be used to estimate the overall severity of the patient's condition. The score ranges from 0 to 4, with higher scores indicating more severe conditions.

SECONDARY OUTCOMES:
erythema index | 0,3,7,14,30,60 days
  Use non-invasive skin analyzer to measure the erythema index on the patient's facial skin at each follow-up visit.The larger the value, the more severe the erythema.
melanin index | 0,3,7,14,30,60 days
  Use non-invasive skin analyzer to measure the melanin index on the patient's facial skin at each follow-up visit.The larger the value, the higher the melanin level.
transepidermal water loss | 0,3,7,14,30,60 days
  Use non-invasive skin analyzer to measure the transepidermal water loss on the patient's facial skin at each follow-up visit.The larger the value, the more severe the transdermal water loss.
hydration | 0,3,7,14,30,60 days
  Use non-invasive skin analyzer to measure the hydration on the patient's facial skin at each follow-up visit.The larger the value, the more severe the hydration.
ECCA score | 0,60 days
GAGS score | 0,60 days
GAIS score | 60 days
Patient satisfaction evaluation | 60 days
  Patient satisfaction was evaluated as very satisfied, satisfied, relatively satisfied and dissatisfied.

CONTACTS AND LOCATIONS:
Locations (1):
- 1927-Nm Fractional Thulium Fiber Laser, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No